CLINICAL TRIAL: NCT04407611
Title: Testing Scalable Communication Modalities for Returning Breast Cancer Genetic Research Results to African American Women
Brief Title: Scalable Communication Modalities for Returning Genetic Research Results
Acronym: BWHS RoR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University of Washington (Other); MGH Institute of Health Professions (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-40045; R01MD014312 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-05-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Breast and Ovarian Cancer; Lynch Syndrome
Keywords: BRCA testing; Return of genetic research results; eHealth; Digital health; Risk communication; ELSI
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Intervention Model Description: Randomization to 1 of 2 study arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional modality (No Intervention): Control arm. Conventional modality entails telephone disclosure of genetic results by a licensed genetic counselor.
- Online modality (Experimental): Online self-guided modality entails return of genetic results directly to participants, with optional genetic counselor follow-up via telephone.
  Interventions: Behavioral: Online modality; Behavioral: Genetic counselor follow-up

INTERVENTIONS:
Behavioral: Online modality — Return of BRCA results directly online or return of printed BRCA results if participant cannot access online or chooses not to
  Other Names: Web modality
  Arms: Online modality
Behavioral: Genetic counselor follow-up — Optional genetic counselor follow-up over the telephone
  Arms: Online modality

SUMMARY:
Efforts to examine the utility of alternate modalities for genetic results disclosure has widespread implications for how precision medicine research might yield direct health benefits for study participants. This study will examine the efficacy of an online self-guided program to return genetic results to a racial minority cohort population. Study results will provide empirical evidence on the effectiveness of alternate modalities for genetic results return, inform ongoing efforts to establish scalable approaches for effective return of genetic research results, and increase access to personal health information among African American women.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) within the Black Women's Health Study (BWHS) to test alternate communication modalities for results disclosure. The BWHS is an ongoing prospective cohort study of 59,000 self-identified black women from across the United States who have been followed since 1995. Targeted sequencing of over 4000 women within the cohort for BRCA1/2 and other known or suspected high and moderate penetrance genes opens up the possibility of returning breast cancer genetic results to BWHS participants and examining the clinical utility of genetic results return. The primary aim of the proposed research project is to compare the efficacy of two communication modalities for returning breast cancer genetic research results to African American women: 1) a conventional modality that entails telephone disclosure by a licensed genetic counselor, and 2) an online self-guided modality that entails returning results directly to participants, with optional genetic counselor follow-up via telephone. Secondary aims of this study will examine 1) moderators of the intervention impact and 2) psychosocial, sociodemographic, and clinical predictors of result uptake. This study is uniquely situated to provide critical empirical evidence on the effectiveness of alternate models for genetic results return and provide further insight into the factors influencing uptake of genetic information among African American women.

ELIGIBILITY:
Inclusion Criteria:

-Women in the BWHS previously included in the targeted breast cancer sequencing project

Exclusion Criteria:

* Women with known cognitive impairments
* Women with variant of uncertain significance (VUS) results from the sequencing study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 932 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participant that decide to learn genetic results at 6 weeks | 6 weeks
  Decisions about learning genetic results for hereditary breast and ovarian cancer will be monitored and recorded in the electronic study database system.
Number of participant that decide to learn genetic results at 6 months | 6 months
  Decisions about learning genetic results for hereditary breast and ovarian cancer will be monitored and recorded in the electronic study database system.
Change from baseline in breast cancer genetics knowledge based on questionnaire at responses at 6 weeks | Baseline, 6 weeks
  Knowledge about breast cancer genetics will be assessed using an investigator derived questionnaire consisting of 16 items. Higher scores out of ten are associated with more genetics knowledge.
Change in baseline depression at 6 weeks | Baseline, 6 weeks
  Depression will be assessed using the the 2-item Patient Health Questionnaire (PHQ-2). The 2 questions are: Over the past 2 weeks have you been bothered by: (1) Little interest or pleasure in doing things, and (2) Feeling down, depressed or hopeless. Responses range from 0 to 3 where 0=Not at all, to 3=Nearly everyday. Scores are added and can range from 0 to 6, with higher scores reflecting greater depression.
Depression at 6 months | 6 months
  Depression will be assessed using the the 2-item Patient Health Questionnaire (PHQ-2). The 2 questions are: Over the past 2 weeks have you been bothered by: (1) Little interest or pleasure in doing things, and (2) Feeling down, depressed or hopeless. Responses range from 0 to 3 where 0=Not at all, to 3=Nearly everyday. Scores are added and can range from 0 to 6, with higher scores reflecting greater depression.
Depression at 12 months | 12 months
  Depression will be assessed using the the 2-item Patient Health Questionnaire (PHQ-2). The 2 questions are: Over the past 2 weeks have you been bothered by: (1) Little interest or pleasure in doing things, and (2) Feeling down, depressed or hopeless. Responses range from 0 to 3 where 0=Not at all, to 3=Nearly everyday. Scores are added and can range from 0 to 6, with higher scores reflecting greater depression.
Change in baseline anxiety at 6 weeks | Baseline, 6 weeks
  Anxiety will be assessed using the the 2-item Generalized Anxiety Disorder scale (GAD-2). The 2 questions are: Over the past 2 weeks how often have you been bothered by the following problems: (1) Feeling nervous, anxious or on edge, and (2) Not being able to stop or control worrying. Responses range from 0 to 3 where 0=Not at all, to 3=Nearly everyday. Scores are added and can range from 0 to 6, with higher scores reflecting greater anxiety.
Anxiety at 6 months | 6 months
  Anxiety will be assessed using the the 2-item Generalized Anxiety Disorder scale (GAD-2). The 2 questions are: Over the past 2 weeks how often have you been bothered by the following problems: (1) Feeling nervous, anxious or on edge, and (2) Not being able to stop or control worrying. Responses range from 0 to 3 where 0=Not at all, to 3=Nearly everyday. Scores are added and can range from 0 to 6, with higher scores reflecting greater anxiety.
Anxiety at 12 months | 12 months
  Anxiety will be assessed using the the 2-item Generalized Anxiety Disorder scale (GAD-2). The 2 questions are: Over the past 2 weeks how often have you been bothered by the following problems: (1) Feeling nervous, anxious or on edge, and (2) Not being able to stop or control worrying. Responses range from 0 to 3 where 0=Not at all, to 3=Nearly everyday. Scores are added and can range from 0 to 6, with higher scores reflecting greater anxiety.
Participant distress from cancer risk assessment (test-specific distress) at 6 weeks | 6 weeks
  Using the Multidimensional Impact of Cancer Risk Assessment (MICRA) distress subscale, the investigators will assess perceptions of distress resulting from learning genetic test results. The distress subscale has 6 items, each scored on a 4 point scale, with higher scores reflecting greater distress.
Participant distress from cancer risk assessment (test-specific distress) at 6 months | 6 months
  Using the Multidimensional Impact of Cancer Risk Assessment (MICRA) distress subscale, the investigators will assess perceptions of distress resulting from learning genetic test results. The distress subscale has 6 items, each scored on a 4 point scale, with higher scores reflecting greater distress.
Participant distress from cancer risk assessment (test-specific distress) at 12 months | 12 months
  Using the Multidimensional Impact of Cancer Risk Assessment (MICRA) distress subscale, the investigators will assess perceptions of distress resulting from learning genetic test results. The distress subscale has 6 items, each scored on a 4 point scale, with higher scores reflecting greater distress.
Participant uncertainty from cancer risk assessment at 6 weeks | 6 weeks
  Using the Multidimensional Impact of Cancer Risk Assessment (MICRA) uncertainty subscale, the investigators will assess perceptions of uncertainty resulting from learning genetic test results. Then uncertainty subscale has 9 items, each scored on a 4 point scale, with higher scores reflecting greater uncertainty.
Participant uncertainty from cancer risk assessment at 6 months | 6 months
  Using the Multidimensional Impact of Cancer Risk Assessment (MICRA) uncertainty subscale, the investigators will assess perceptions of uncertainty resulting from learning genetic test results. Then uncertainty subscale has 9 items, each scored on a 4 point scale, with higher scores reflecting greater uncertainty.
Participant uncertainty from cancer risk assessment at 12 months | 12 months
  Using the Multidimensional Impact of Cancer Risk Assessment (MICRA) uncertainty subscale, the investigators will assess perceptions of uncertainty resulting from learning genetic test results. Then uncertainty subscale has 9 items, each scored on a 4 point scale, with higher scores reflecting greater uncertainty.

CONTACTS AND LOCATIONS:
Overall Officials: Catharine Wang, PhD, Principal Investigator — BU School of Public Health
Locations (1):
- BU School of Public Health, the research is being conducted remotely, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Bertrand KA, Trevino-Talbot M, Flynn M, Ruderman M, Cabral HJ, Bowen DJ, Hughes-Halbert C, Palmer JR. Ethical, legal, and social implications (ELSI) and challenges in the design of a randomized controlled trial to test the online return of cancer genetic research results to U.S. Black women. Contemp Clin Trials. 2023 Sep;132:107309. doi: 10.1016/j.cct.2023.107309. Epub 2023 Jul 27. PMID 37516165

DOCUMENTS (1):
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT04407611/ICF_000.pdf